CLINICAL TRIAL: NCT00743990
Title: Effect of a Medicated Topical Therapy, Petrolatum, and No Treatment on Nocturnal Cough and Congestion for Children With Upper Respiratory Infections
Brief Title: Effect of Effect of a Medicated Topical Therapy , Petrolatum, and No Treatment on Nocturnal Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29273
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Respiratory Tract Diseases
Keywords: Cough symptoms; Cold symptoms; Congestion; Children; URI; Alternative cough symptom treatment
MeSH Terms: conditions — Respiratory Tract Diseases; Cough | interventions — Eucalyptus Oil; Menthol; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator)
  Interventions: Other: Ointment containing camphor, eucalyptus oil, and menthol
- B (Placebo Comparator)
  Interventions: Other: Petroleum jelly
- 3 (No Intervention): no intervention

INTERVENTIONS:
Other: Ointment containing camphor, eucalyptus oil, and menthol — One time use
  Arms: A
Other: Petroleum jelly — One time use
  Arms: B

SUMMARY:
This study seeks to subjectively evaluate whether a single application of Vicks® VapoRub® (VVR) ointment or a control ointment (petrolatum) will be superior to no treatment for control of nocturnal cough and congestion due to upper respiratory tract infection (URI) as rated by both parents and children.

ELIGIBILITY:
Inclusion Criteria:

* Cough and congestion attributed to upper respiratory tract infection

Exclusion Criteria:

* Children with signs or symptoms of more serious or treatable disease
* Presence of itchy, watery eyes or frequent sneezing
* Tachypnea (respiratory rate >95%ile) or labored breathing
* Symptoms for 8 or more days
* History of asthma in the past 2 years, chronic lung disease, or seizure disorder
* History of an allergic reaction to camphor, menthol, eucalyptus, petrolatum, cedarleaf oil, nutmeg oil, thymol, turpentine oil, Over-the-counter medication containing VVR components

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Subjective assessment of cough and congestion symptoms | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Paul, MD, MSc, Principal Investigator — Penn State University
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Paul IM, Beiler JS, King TS, Clapp ER, Vallati J, Berlin CM Jr. Vapor rub, petrolatum, and no treatment for children with nocturnal cough and cold symptoms. Pediatrics. 2010 Dec;126(6):1092-9. doi: 10.1542/peds.2010-1601. Epub 2010 Nov 8. PMID 21059712